CLINICAL TRIAL: NCT01384526
Title: Investigating the Impact of Tamoxifen Therapy on Ovarian Aging
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 025950
Record Dates: First submitted 2011-06-24; First posted 2011-06-29 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Fertility
Keywords: hormone therapy; ovarian aging; ovarian reserve; fertility; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum AMH, FSH, estradiol, and Inhibin B will be measured. Blood will be collected and processed by the UCSF Center for Reproductive Health. Serum samples will be stored at -80oC in a designated freezer with an alarm system. Biomarker assessments will be performed by Quest Laboratories under standard quality control.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- history of hormone therapy
- no history of hormone therapy

SUMMARY:
Ovarian toxicity is a well-described side effect of traditional chemotherapy in premenopausal women receiving treatment for early stage breast cancer. However, the impact of long-term endocrine therapy on ovarian function is not established, and to our knowledge, has never been directly studied. Understanding the effects of hormone therapy on ovarian aging will help breast cancer patients of reproductive age make more informed and empowered decisions regarding their treatment. The purpose of this study is to explore the relationship between tamoxifen therapy and ovarian aging. Patients will be identified through the UCSF Cancer Registry and California Pacific Medical Center Cancer Registry and will be evaluated based on age and menopausal status. Women who read about the study from clinicaltrials.gov and contact the study coordinator will also be considered for enrollment. The age of menopause onset will be assessed through surveys and will be compared to the accepted national average age of natural menopause. Biomarkers of ovarian reserve will be assessed in premenopausal women between ages 25-45 and will be compared to those of healthy age- and ethnicity-matched premenopausal controls from an ongoing RO1- funded prospective longitudinal ovarian aging (OVA) study.

ELIGIBILITY:
Inclusion Criteria

1. Female
2. ≥25 years of age at the time of study enrollment
3. Diagnosed with stage I-III invasive breast cancer or ductal carcinoma in situ, or determined to be high risk for primary breast cancer
4. If endocrine therapy was used, women must have completed at least 2 years of endocrine therapy as defined by either

   1. Tamoxifen alone
   2. Ovarian suppression plus tamoxifen or aromatase inhibitor
   3. Ovarian suppression alone
5. Women must have been premenopausal at the time of endocrine therapy initiation. Premenopausal is defined as having had a menstrual cycle within 12 months before starting treatment.
6. For the biomarker assessments, patients must be off all endocrine therapy (tamoxifen, ovarian suppression with goserelin or leuprolide, or aromatase inhibitor) for at least 6 months prior to study enrollment.
7. For the biomarker assessments, patient must be off hormone contraceptives, fertility treatments, or other hormone therapies for at least 3 months prior to study enrollment
8. For the biomarker assessments, patient must have had regular periods the last 3 months.

Exclusion Criteria

1. Evidence for either local recurrence following use of adjuvant systemic therapy or evidence for distant recurrence of breast cancer.
2. Prior history of ovarian surgery or manipulation
3. Mother with premature ovarian failure as defined by onset of menopause at age <40
4. Prior chemotherapy exposure
5. Prior history of endometriosis, anovulation or documented infertility
6. Pregnant at the time of study enrollment

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The UCSF Cancer Registry will be screened for female patients who were treated at the UCSF Breast Care Center between 1985 and 2010 and who meet the eligibility criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
age of menopause onset | assessed at time of reproductive history survey (30 minutes long, one-time assessment)
  The primary aim of this study is to determine the mean age of menopause onset in a cohort of women who have completed a course of tamoxifen therapy and to compare this age with the accepted national average age of natural menopause. Age of menopause onset which is defined as the year of the last menstrual period minus patient's birth year.

SECONDARY OUTCOMES:
biomarkers of ovarian reserve | assessed at time of ultrasound and blood draw (single day appointment, 1 hour)
  A secondary aim is to compare biomarkers of ovarian reserve in premenopausal women between ages 25-45 who have been previously treated with tamoxifen with those of age- and ethnicity-matched healthy controls. The primary biomarker of interest is antral follicle count (AFC). Other biomarkers that will be measured include anti-Mullerian hormone (AMH), inhibin B, FSH, and estradiol levels.
reproductive history | assessed at time of reproductive history survey (30 minutes long, one-time assessment)
  A secondary aim is to characterize the reproductive histories of women who have completed a course of endocrine therapy for the prevention or treatment of breast cancer.
lifestyle factors, medical history, and demographics | assessed at time of reproductive history survey (30 minutes long, one-time assessment)
  A secondary aim is to correlate biomarkers of ovarian age and age of menopause onset with lifestyle factors, medical history, and demographics in pre- and postmenopausal women previously treated with endocrine therapy, accounting for age and ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: A. Jo Chien, MD, Principal Investigator — University of California, San Francisco; Mitch Rosen, MD, Principal Investigator — UCSF Center for Reproductive Health
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States